CLINICAL TRIAL: NCT04522986
Title: An Exploratory Study of ADR-001 in Patients with Severe Pneumonia Caused by SARS-CoV-2 Infection
Acronym: COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rohto Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADR-001-1919
Record Dates: First submitted 2020-08-20; First posted 2020-08-21 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mesenchymal stem cell (Experimental): 4 times dose of Mesenchymal stem cell
  Interventions: Biological: Mesenchymal stem cell

INTERVENTIONS:
Biological: Mesenchymal stem cell — 1*10^8 cells are administered once a week, total four times intravenously.

SUMMARY:
Safety and efficacy of ADR-001 are evaluated in Patients with Severe Pneumonia caused by SARS-CoV-2 infection.

DETAILED DESCRIPTION:
Patients with Severe Pneumonia caused by SARS-CoV-2 infection are enrolled to the study. Adipose-derived mesenchymal stem cells (AD-MSCs) are administered once a week, total four times intravenously. Safety and efficacy of AD-MSCs are evaluated for 12 weeks after first administer.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 infection is confirmed on antigen test or PCR test
* Pulmonary infiltrative shadow is confirmed on chest X-ray test
* Mechanical ventilation is being utilized, or Acute Respiratory Failure whose PaO2 is not being achieved to 80 mmHg in spite of High-flow oxygen therapy

Exclusion Criteria:

* Continue treatment for Pneumonia before SARS-CoV-2 infection
* SOFA score >= 15
* Infection type on DIC diagnosis criteria >= 4
* Deep Venous Thrombosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Safety: Adverse Event | 12 weeks
  Adverse events which appear in subjects with ADR-001 treatment are evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Yuji Fujino, MD, Principal Investigator — Osaka University Hospital
Locations (1):
- Osaka University Hospital, Suita, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No